CLINICAL TRIAL: NCT06295419
Title: Comparison of the Effect of Dual Task on Manual Ability Performance in Children With Cerebral Palsy With Healthy Controls
Brief Title: The Effect of Dual Task on Manual Ability Performance in Children With Cerebral Palsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Igdir University (Other)
Responsible Party: Principal Investigator, Sema Bugusan Oruc, Head of Physiotherapy and Rehabilitation Department, Igdir University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Igdir182
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Cerebral Palsy
Keywords: cerebral Palsy; dual-task; manual ability; trunk control
MeSH Terms: conditions — Cerebral Palsy | interventions — potassium channel subfamily K member 3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cerebral palsy (Experimental): cerebral palsy will be evaluated single and dual task conditions
  Interventions: Other: dual task; Other: single task
- healthy controls (Experimental): Healthy controls will be evaluated single and dual task conditions
  Interventions: Other: dual task; Other: single task

INTERVENTIONS:
Other: dual task — cerebral palsy and healthy controls will be evaluated dual task conditions
Other: single task — cerebral palsy and healthy controls will be evaluated single task conditions

SUMMARY:
The aim of the study is to investigate the effect of dual task conditions on manual dexterity performance in young people and children with CP between the ages of 7-18 and to compare it with their peers.

Evaluations to be made in the study (children with CP) and control (typically developing peers) groups:

* Demographic information, Gross Motor Function Level (GMFCS), Manual Skills Classification System (MACS) and dominant extremity will be noted and the evaluation will begin by applying the Abilhand Kids questionnaire.
* Firstly, the child's performance on a single cognitive task will be evaluated in a supported sitting position on a chair. The cognitive task will be the n-back task (counting down task) to be applied in accordance with the level of the child or young person.
* Using the Visual Analogue Scale (VAS), participants will be asked to score the difficulty of the cognitive task as a number between 0 and 10.
* In order to evaluate the single motor performance of manual skills, the 9-Hole Test will be applied and the times will be recorded by asking to write a given paragraph.
* Dual task evaluations will be administered by giving a simultaneous cognitive task while administering the 9-Hole Test and writing a paragraph.
* In order to reveal the dual-task cost (DTC), dual-task performance will be subtracted from single-task performance and the difference will be calculated in seconds.
* The Body Control Measurement Scale will be applied for body evaluation purposes.

As a result of this study, the changes in manual dexterity and cognitive performance in dual-task conditions in children and adolescents with CP will be revealed. Additionally, changes in this performance in dual-task situations will be compared with a control group of typically developing children.

DETAILED DESCRIPTION:
In the literature, balance or walking postural tasks are mostly used in dual-task studies for children and young people with Cerebral Palsy (CP). However, dual task tasks performed during manual skills in daily life have not been adequately researched. The aim of the study is to investigate the effect of dual task conditions on manual dexterity performance in young people and children with CP between the ages of 7-18 and to compare it with their peers. Although studies on this subject in the world are limited.

MATERIAL AND METHOD:

Evaluations to be made in the study (children with CP) and control (typically developing peers) groups:

-Demographic information, Gross Motor Function Level (GMFCS), Manual Skills Classification System (MACS) and dominant extremity will be noted and the evaluation will begin by applying the Abilhand Kids questionnaire.

Abilhand Kids is a questionnaire that evaluates children's upper extremities bimanually, has proven validity and reliability, and includes 21 questions for families about the common tasks their children undertake in daily life activities.

* Firstly, the child's performance on a single cognitive task will be evaluated in a supported sitting position on a chair. The cognitive task will be the n-back task (counting down task) to be applied in accordance with the level of the child or young person.
* Using the Visual Analogue Scale (VAS), participants will be asked to score the difficulty of the cognitive task as a number between 0 and 10.
* In order to evaluate the single motor performance of manual skills, the 9-Hole Test will be applied and the times will be recorded by asking to write a given paragraph.
* Dual task evaluations will be administered by giving a simultaneous cognitive task while administering the 9-Hole Test and writing a paragraph.
* In order to reveal the dual-task cost (DTC), dual-task performance will be subtracted from single-task performance and the difference will be calculated in seconds.
* The Body Control Measurement Scale will be applied for body evaluation purposes.

The scale consists of 15 items in total (subscales 5, 7 and 3 items, respectively). Items are scored on an ordinal scale of 2, 3, and 4 points. Although the total score of the scale varies between 0-58 points, higher scores indicate better performance. The Turkish validity and reliability of the survey was conducted.

As a result of this study, the changes in manual dexterity and cognitive performance in dual-task conditions in children and adolescents with CP will be revealed. Additionally, changes in this performance in dual-task situations will be compared with a control group of typically developing children.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 7-15,
* Not having a chronic disease.

Exclusion Criteria:

* Participants must have had Botulinum Toxin applied to the upper extremity in the last 6 months
* Participants must have had a health problem or had an operation that would affect the musculoskeletal system or dexterity performance in the last year (EX: Distal radius fracture).
* Having concentration problems such as attention deficit hyperactivity disorder (ADHD).
* Not volunteering to participate in the study and not signing a consent form.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Abilhand Kids | 5minutes
  Abilhand Kids is a questionnaire that evaluates children's upper extremities bimanually, has proven validity and reliability, and includes 21 questions for families about the common tasks their children undertake in daily life activities.
cognitive task (single task) | 1minute
  The cognitive task will be the n-back task (counting down task) to be applied in accordance with the level of the child or young person.
motor performance of manual skills (writing a paragraph) (single task) | 2minutes
  the time will be recorded by asking to write a given paragraph.
motor performance of manual skills (single task) | 2minutes
  the 9-Hole Peg Test will be applied and the time will be recorded.
motor performance of manual skills (dual task) | 2minutes
  Dual task evaluations will be administered by giving a simultaneous cognitive task while administering the 9-Hole Peg Test. And the time will be recorded.
motor performance of manual skills (writing a paragraph) (dual task) | 2minutes
  Dual task evaluations will be administered by giving a simultaneous cognitive task while writing a paragraph. And the time will be recorded.
The Body Control Measurement Scale | 10minutes
  The scale consists of 15 items in total (subscales 5, 7 and 3 items, respectively). Items are scored on an ordinal scale of 2, 3, and 4 points. Although the total score of the scale varies between 0-58 points, higher scores indicate better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Sema Büğüşan Oruç, PhD, Principal Investigator — Igdir University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reilly DS, Woollacott MH, van Donkelaar P, Saavedra S. The interaction between executive attention and postural control in dual-task conditions: children with cerebral palsy. Arch Phys Med Rehabil. 2008 May;89(5):834-42. doi: 10.1016/j.apmr.2007.10.023. PMID 18452729
- [Background] Gathercole SE, Pickering SJ, Ambridge B, Wearing H. The structure of working memory from 4 to 15 years of age. Dev Psychol. 2004 Mar;40(2):177-90. doi: 10.1037/0012-1649.40.2.177. PMID 14979759
- [Background] Pena GM, Pavao SL, Oliveira MF, de Campos AC, Rocha NA. Dual-task effects in children with neuromotor dysfunction: a systematic review. Eur J Phys Rehabil Med. 2019 Apr;55(2):281-290. doi: 10.23736/S1973-9087.19.05556-4. Epub 2019 Jan 8. PMID 30621370
- [Background] Wollesen B, Janssen TI, Muller H, Voelcker-Rehage C. Effects of cognitive-motor dual task training on cognitive and physical performance in healthy children and adolescents: A scoping review. Acta Psychol (Amst). 2022 Apr;224:103498. doi: 10.1016/j.actpsy.2022.103498. Epub 2022 Jan 25. PMID 35091209
- [Background] Rubsam M, Girolami GL, Bhatt T. Heterogeneity of Tasks and Outcome Measures in Dual Tasking Studies in Children With Cerebral Palsy: A Scoping Review. Phys Ther. 2024 Jan 1;104(1):pzad151. doi: 10.1093/ptj/pzad151. PMID 37941469